CLINICAL TRIAL: NCT03937401
Title: Use of Oxytocin in MRI-HIFU Treatment
Brief Title: Oxytocin in MRI-HIFU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T366/2017
Record Dates: First submitted 2019-04-26; First posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Fibroid; Adenomyosis
Keywords: oxytocin; MRI-HIFU; fibroid; adenomyosis
MeSH Terms: conditions — Leiomyoma; Adenomyosis | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients treated with oxytocin during MRI-HIFU (Experimental)
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin infusion during MRI-HIFU treatment
  Other Names: MRI-HIFU

SUMMARY:
Capability of oxytocin in improving the efficacy of MRI-HIFU is studied. Patients undergoing MRI-HIFU treatment are given oxytocin during treatment and the efficacy of the treatment will be analysed by patient reported symptom questionnaires and imaging data.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing MRI-HIFU -treatment
* Patients assessed for suitability to MRI-HIFU treatment
* willingness to participate in trial

Exclusion Criteria:

* Known allergy to Syntocinon/oxytocin
* Elevated blood pressure
* ischemic heart disease
* Long QT- interval

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
NPV | up to one year
  non perfused volume (percentage of fibroid destroyed)
duration of MRI-HIFU | up to one year
  duration of MRI-HIFU treatment
UFS-Qol | 12 months after HIFU treatment
  Uterine fibroid symptom severity and quality of life (patient quality of life questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers

REFERENCES:
- [Derived] Otonkoski S, Viitala A, Komar G, Sainio T, Yanovskiy A, Blanco Sequieros R, Perheentupa A, Joronen K. Magnetic resonance guided high intensity focused ultrasound (MR-HIFU) effectively reduces fibroid-related symptoms and improves quality of life-A prospective single-centre 12-month follow-up study. Acta Obstet Gynecol Scand. 2025 Jun;104(6):1172-1180. doi: 10.1111/aogs.15086. Epub 2025 Apr 29. PMID 40302212
- [Derived] Otonkoski S, Sainio T, Komar G, Suomi V, Saunavaara J, Blanco Sequeiros R, Perheentupa A, Joronen K. Oxytocin selectively reduces blood flow in uterine fibroids without an effect on myometrial blood flow: a dynamic contrast enhanced MRI evaluation. Int J Hyperthermia. 2020;37(1):1293-1300. doi: 10.1080/02656736.2020.1846792. PMID 33207939